CLINICAL TRIAL: NCT02328703
Title: Reiki for the Management of Neuropathic Pain in Service Members With Extremity Trauma
Brief Title: Reiki for the Management of Neuropathic Pain
Acronym: Reiki4Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to substantial decrease in the desired patient population.
Sponsor: Fort Belvoir Community Hospital (U.S. Federal Agency)
Collaborators: Defense and Veterans Center for Integrative Pain Management (Other); University of Pennsylvania (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, LTC MeLisa Gantt, (former) Chief, Research Programs, Fort Belvoir Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 375746; N12-P10 (Other Grant/Funding Number: TriService Nursing Research Program)
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Neuropathic Pain; Amputation, Traumatic
Keywords: Reiki; Neuropathic Pain; Military Service Members; Extermity Trauma
MeSH Terms: conditions — Neuralgia; Amputation, Traumatic | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reiki Therapy by a Reiki Master (Experimental): The Reiki Master will take approximately 30 minutes to perform a hand placement sequence that will allow the direction of energy toward the site of pain.
  Interventions: Other: Reiki Therapy
- Sham Reiki Therapy by a Clinician (Placebo Comparator): The Clinician, who has not trained in Reiki, will mimic the same 30 minute hand placement protocol as the Reiki Master.
  Interventions: Other: Reiki Therapy

INTERVENTIONS:
Other: Reiki Therapy — Reiki is a biofield energy therapy that is based on the idea that there is a universal energy that supports the body's innate healing abilities. A trained Reiki Master uses their hands as a conduit of the energy that goes naturally to any area of the recipient's body where it is needed. This provides a means for life force energy to recharge and rebalance the human energy fields, creating optimal conditions needed by the body's natural healing system.

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled, repeated measures study with intention-to-treat that involves exposure to Reiki therapy or a placebo control intervention for a total of six treatments, three treatments per week for two weeks, with a 2-week follow-up for the decrease of neuropathic pain in extremity trauma.

DETAILED DESCRIPTION:
Sixty participants will be randomized to either receive three 30-minute standardized treatments per week for two weeks of Reiki therapy (n=30) or a placebo intervention (n=30). All participants will complete the same outcome measures (Brief Pain Inventory, Neuropathic Pain Scale, Patient Global Impression of Improvement Scale, Pittsburgh Quality of Sleep Scale, and McGill Pain Questionnaire-SF) at established times. Any opioid and other analgesic requirements will also be collected.

Aim 1: Test the efficacy of a 2-week course of Reiki therapy on pain outcomes (present, average and worst pain intensity levels and perceptions of pain relief from the Brief Pain Inventory (BPI) and Patient Global Impression of Improvement-PGI-I) compared to placebo Reiki interventions in combat-injured service members with major limb trauma experiencing neuropathic pain.

Aim 2: Examine effects of a 2-week course of Reiki therapy compared to placebo Reiki interventions on the quality of sleep measured by the Pittsburgh Sleep Quality Index (PSQI), pain interference (BPI), character and quality of pain (Neuropathic Pain Scale and McGill Pain Questionnaire-Short Form) in combat-injured service members with major limb trauma experiencing neuropathic pain.

Aim 3: Describe the differences in pattern of responses to Reiki therapy and placebo Reiki interventions for pain outcomes (pain intensity, perception of relief and PGI-I) based on neuropathic pain type, pain duration, and the presence or absence of a diagnosis of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Be Active, Reserve, or National Guard with previous deployment(s) to OIF, OEF, or OND
* Be age 18 years or older
* Have ability to read and understand consent forms and study documents
* Have sustained at least one traumatic combat extremity injury defined as: single or both arm or leg, above or below knee amputation, mangled limb(s)
* Report, from a major traumatic extremity injury, an average and worst pain level ≥ 5 (numeric rating scale of 0 to 10) for at least one of three days prior to enrollment
* Be receiving a stable pain medication regimen defined as a regimen that may include multimodal analgesia with opioids, anticonvulsants and/or antidepressants for neuropathic pain in relatively stable doses with no more than a 10 to 20% increase over the past week prior to enrollment
* Have a cognitive performance evaluation that is consistent with an understanding of the proposed study as assessed by a "teach back" process
* Be receiving a minimum of two hours of physical therapy per day

Exclusion Criteria:

* Moderate to severe traumatic brain injury (TBI) as documented on the standardized evaluation completed by TBI Service providers
* Active moderate to severe psychological distress or psychiatric condition such as active psychosis, suicidal or homicidal ideation as documented, on the standardized psychological evaluation completed by a behavioral health psychiatrist
* Pregnancy
* Any medical condition that in the opinion of the participant's health care provider or PI has the potential to interfere with the effects of Reiki treatments
* Being pre-scheduled for additional surgeries or major painful and activity limiting procedures during the participant's participation in the study
* Received Reiki therapy treatment within the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Participants will be followed from start of treatment to up to 4 weeks
  The BPI Short Form assesses the time relation sensory component of pain intensity (average over the last week, worst and least, and present pain) using a numeric rating scale (0 [No pain] to 10 [Pain as bad as you can imagine]), percentage of pain relief (0 [No relief] to 100% [Complete relief]), and 7 pain interferences concerning work, activity, mood, enjoyment, sleep, walk and relationships are assessed using 0-10 numeric scales (0 [No interference] to 10 [Complete interference])
Neuropathic Pain Scale (NPS) | Participants will be followed from start of treatment to up to 4 weeks
  The NPS assesses two pain domains (intensity and unpleasantness), six qualities (sharp, hot, dull, cold, sensitive, and itchy) and two locations (deep and surface).
McGill Pain Questionnaire-Short Form (MPQ-SF) | Participants will be followed from start of treatment to up to 4 weeks
  The MPQ-SF is a brief screening tool for pain and has 3 subscales: Sensory (11 word items), Affective (4 word items), and a composite Evaluative score. Fifteen words represent acute, intermittent and chronic pains, and are scored on a four-point Likert-type scale from 0 = none to 3 = severe. A total score of 45 is possible by summing the Sensory and Affective subscales and scoring them separately.
Pittsburgh Sleep Quality Index (PSQI) | Participants will be followed from start of treatment to up to 4 weeks
  The PSQI assesses sleep quality and disturbances over a 1-month time interval will be evaluated using the PSQI (Appendix J). Nineteen items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and day time dysfunction. The sum of scores yields one global score.
Patient Global Impression of Improvement Scale (PGI-I) | Participants will be followed from start of treatment to up to 4 weeks
  The PGI-I consists of a 7-point Likert scale with 1 = "very much improved" to 7 = "very much worse" to capture overall changes related to a study medication or intervention

CONTACTS AND LOCATIONS:
Overall Officials: MeLisa Gantt, PhD, Principal Investigator — Fort Belvoir Community Hospital
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States